CLINICAL TRIAL: NCT05447767
Title: Prediction AlgoriThm for regeneraTive Medicine Approach in knEe OA: New Decision-making Process Based on Patient pRofiliNg. (CO-2019-12370720 Prof. Kon BANDO DI RICERCA FINALIZZATA 2019)
Brief Title: Prediction AlgoriThm for regeneraTive Medicine Approach in knEe OA: New Decision-making Process Based on Patient pRofiliNg (PATTERN)
Acronym: PATTERN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Ministero della Salute, Italy (Other); Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2921
Record Dates: First submitted 2022-03-25; First posted 2022-07-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- intra-articular injection of BMAC (Active Comparator): intra-articular injection of BMAC
  Interventions: Device: KIT BMAC
- intra-osseous and intra-articular injection of BMAC (Active Comparator): intra-osseous and intra-articular injection of BMAC
  Interventions: Device: KIT BMAC
- intra-articular injection of at- SVF (Active Comparator): intra-articular injection of at- SVF
  Interventions: Device: at-SVF FIDIA
- intraosseous and intra-articular injection of at-SVF (Active Comparator): intraosseous and intra-articular injection of at-SVF
  Interventions: Device: at-SVF FIDIA

INTERVENTIONS:
Device: KIT BMAC — intra-articular infiltration of BMAC
  Arms: intra-articular injection of BMAC
Device: KIT BMAC — intra-articular and intra-osseous infiltration of BMAC
  Arms: intra-osseous and intra-articular injection of BMAC
Device: at-SVF FIDIA — intra-articular infiltration of at-SVF
  Arms: intra-articular injection of at- SVF
Device: at-SVF FIDIA — intra-articular and intra-osseous infiltration of at-SVF
  Arms: intraosseous and intra-articular injection of at-SVF

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease characterised by chronic pain, degradation and loss of articular cartilage, osteophyte formation and varying degrees of synovial inflammation.

Today, most of the available conservative treatments provide temporary relief of symptoms but have no effect on the cause and progression of the disease. Mesenchymal stem cells (MSC) have emerged as a durable and effective conservative treatment option for OA.

They are tissue cell-rich concentrates that have demonstrated immunomodulatory activities in several in vitro and in vivo studies, particularly in orthopaedics.

Thus, "minimal handling" methods for the intraoperative production of tissue cell-rich concentrates has become a widespread strategy in clinical practice. In particular, bone marrow aspirate concentrate (BMAC) and adipose tissue enriched SVF (at-SVF), i.e. the so-called 'orthobiologics', have proven to be cost-effective and promising sources with a high safety profile and positive short-term clinical results.

Despite growing evidence on the use of orthobiologics, the different methods of preparation and administration and the lack of meaningful data collection do not allow for a clear understanding of the true efficacy of these treatments, resulting in a lack of patient-specific indications.

Although the most common method of administering regenerative Although the most common method of administering regenerative medicinal products is by intra-articular injection, more recently it has been shown that in patients with OA the subchondral bone also undergoes significant pathological changes. Given this evidence, intra-osseous (bone-cartilage interface) injections of biological products may represent a promising approach.

DETAILED DESCRIPTION:
Multicentre, open-label, randomised, four-arm clinical trial. Patients enrolled in this clinical trial will undergo scheduled surgery for the treatment of grade 2-3 OA KL. After enrolment, patients will be assigned to 4 treatment groups:

1) intra-articular injection of BMAC, 2) intra-osseous and intra-articular injection of BMAC, 3) intra-articular injection of at-SVF, 4) intra-osseous and intra-articular injection of at-SVF. Medical history, clinical and radiological features, and serum samples will be collected for each patient at baseline, along with cell counts of each product injected.

The primary efficacy objective is the mean change from baseline to 12 months in the mean scores of the Pain and Symptoms in the Knee and Osteoarthritis Outcome Score (KOOS) subscales for each arm.

The KOOS subscale scores of pain and symptoms will be aggregated and averaged as the primary outcome.

Secondary objectives

* Patient profiling through the collection of clinical, radiological and anamnestic data, and through high-throughput proteomic analysis of serum samples and validation of differentially expressed markers to identify possible specific characteristics of responder and non-responder patients to each treatment.
* Whole organ magnetic resonance imaging (WORMS) at 6, 12 months from baseline;
* Presence/appearance of structural pathological features detected by MRI at 6, 12 months compared to baseline;.

This is a post-market clinical investigation of the bone marrow aspirate concentrate (BMAC) and adipose tissue enriched in SVF (at-SVF) for the treatment of OA.

The study is a multicentric, open-label, prospective, 4-arms, in male and female Patients, aged between 18 and 75 years , affected by knee OA Kellgren-Lawrence (KL) 2-3.

The primary objective of this study is to develop an algorithm for the determination of the best treatment for each OA patient, the secondary objective is to identify responder patients to each treatment and to correlate their biologic profile, based on protein expression patterns in the blood samples pre and post-treatment, and the third objective is to compare two autologous bone marrow-derived and adipose-derived treatments on different OA phenotype patients. High-throughput proteomic analysis will be performed on the patients' sera from the 10 top and 10 worst clinical performers in each group at 6 months. Differentially expressed biomarkers will be validated on the whole cohort of patients by commercially available serum tests (ELISA). Data derived from the clinical trial and biomarker assessment will identify all possible covariates influencing the clinical outcome. A principal components analysis will be the base for the development of a prediction algorithm for identification of responders and non-responders to each treatment, in order to provide indications for a personalized approach for knee OA treatment. The markers identified during the high-throughput analysis will be validated using standard diagnostic procedures. A specific diagnostic kit made of reagents and methods for the assessment of the selected and validated biomarkers will be produced and patented. The proteomics analysis on serum samples will be performed at IRCCS Istituto Ortopedico Galeazzi, while markers validation assays will be performed at IRCCS Humanitas.

240 patients affected by knee OA KL 2-3 will enrolled and randomized in 4 treatment groups:

1. intra-articular injection of BMAC;
2. intra-osseous and intra-articular injection of BMAC;
3. intra-articular injection of at- SVF;
4. intraosseous and intra-articular injection of at-SVF. Medical history, clinical and radiological features as well as a serum samples, will be collected for each patient at baseline. Complete cell count will be performed on all injected samples.

Patients will be evaluated at the investigational site for 12 months: at Visit 1 (screening visit, day -90 before treatment), Visit 2 (day of treatment), Visit 3 (Follow-up +3 Months after treatment), Visit 4 (Follow-up +6 Months after treatment), Visit 5 (Follow-up +12 Months after treatment).

Adverse events should be assessed and documented at each scheduled visit starting from signature of informed consent. Adverse events will be evaluated at every visit, with an evaluation of pain and the measurement of health status (quality of life and functional scores); radiological assessments (MRI) will be performed at visit 1, visit 4 and visit 5.

The enrolment will go on until 60 patients are allocated to each group (allocation:1:1:1:1).

Baseline visit/Procedure Visit (V2, Day 0)

During this visit, the investigator will:

1. Review of inclusion/exclusion criteria and confirm patient's eligibility
2. Administer a urine pregnancy test to females of childbearing potential
3. Peripheral blood samples
4. Harvesting Adipose/Bone Tissue preparation with at-SVF/BMAC Kit
5. Injection can be executed under arthroscopical control
6. Record patient's concomitant treatments and medications
7. Record any AEs
8. Cell count of injected products

Follow-up Visit (V3, 3 months ± 4 weeks)

During this visit, the investigator will:

1. Perform physical examination
2. Perform the knee assessment and complete:
3. Administer to the patient the following questionnaires:
4. KOOS subscales
5. IKDC questionnaire
6. VAS score
7. Record patient's concomitant treatments and medications
8. Record any AEs

Follow-up Visit (V4, 6 months ± 6 weeks)

During this visit, the investigator will:

1. Perform physical examination
2. Perform the knee assessment and complete:
3. Administer to the patient the following questionnaires:
4. KOOS subscales
5. IKDC questionnaire
6. Vas Score
7. Administer a urine pregnancy test to females of childbearing potential, before the MR Imaging
8. Submit patient to a MRI
9. Record patient's concomitant treatments and medications
10. Record any AEs

Follow-up Visit (V4, 12 months ± 8 weeks)

During this visit, the investigator will:

1. Perform physical examination
2. Perform the knee assessment and complete:
3. Administer to the patient the following questionnaires:
4. KOOS subscales
5. IKDC questionnaire
6. Vas Score
7. Administer a urine pregnancy test to females of childbearing potential, before the MR Imaging
8. Submit patient to a MRI
9. Record patient's concomitant treatments and medications
10. Record any AEs

In case of premature withdrawal from the study for whatever reason, the same assessments described for Visit 4 will be performed and recorded in an "Early termination visit".

The Investigator will duly record the reason for premature withdrawal in the source documents and then in the appropriate section of the CRF. Visit 4 (12 months ± 8 weeks) or the 'Early termination Visit' will represent the conclusion of patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75;
2. Patients affected by knee OA KL 2-3;
3. Patients understanding the nature of the study and providing their informed consent to participation;
4. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol;
5. Body mass index (BMI) ≤ 40 kg/m2;
6. Ability to provide written informed consent and can understand and comply with the requirements of the study.

Exclusion Criteria:

A 4-arms randomized clinical trial in 240 patients affected by knee OA KL 2-3. Treatment groups: 1) intra-articular injection of BMAC, 2) intra-osseous and intra-articular injection of BMAC, 3) intra-articular injection of adipose tissue enriched in SVF (at-SVF) , 4) intraosseous and intra-articular injection of at-SVF.

Inclusion criteria:

1. Patients aged 18-75;
2. Patients affected by knee OA KL 2-3;
3. Patients understanding the nature of the study and providing their informed consent to participation;
4. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol;
5. Body mass index (BMI) ≤ 40 kg/m2;
6. Ability to provide written informed consent and can understand and comply with the requirements of the study.

Exclusion criteria:

1. Patients with known inflammatory diseases at the time of enrolment.
2. Patients who are not allowed to undergo the study procedures involving imaging (X-rays, MRI) based on Investigator's judgement.
3. A history of local anaesthetic and anticoagulant drug allergy;
4. Clinically observed active infection in the index knee joint or skin disease/breakdown or infection in the area of the planned injection site of the index knee;
5. Major surgery (e.g. osteotomy) of the index knee within 12 months prior to screening;
6. Minor surgery (e.g. shaving or arthroscopy) of the index knee within 6 months prior to screening;
7. Patients who received intra-articular injection of corticosteroids, PRP or HA within the previous 3 months;
8. Use of systemic immunosuppressants within 6 weeks prior to screening;
9. Patients with a history of invasive malignancies (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years;
10. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
11. Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation and for three months later.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
The mean KOOS score change from baseline to 12 months. | 12 months
  KOOS, IKDC and VAS questionnaires will be administered during screening visit and follow-up visits in order to monitor the evolution of the patients. KOOS subscales scores of Pain and Symptoms will be aggregated and averaged as primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05447767/Prot_SAP_000.pdf